CLINICAL TRIAL: NCT03653442
Title: Non-invasive Haemodynamic Parameters Predictive of Hypotension Induced by Neuraxial Anaesthesia During Elective Caesarean Section
Brief Title: Non Invasive Haemodynamics in Neuraxial Anaesthesia Hypotension
Acronym: NIHNAH
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Chiara Viviani, Principal Investigator, Papa Giovanni XXIII Hospital
Other Study IDs: Reg. 2018/0051
Record Dates: First submitted 2018-05-14; First posted 2018-08-31 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Hypotension, Controlled; Anaesthesia, Spinal; Caesarean Section
Keywords: Induced hypotension; Spinal Anaesthesia; Elective Caesarean section; non-invasive haemodynamic parameters
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Spinal (or neuraxial) anaesthesia is still considered the first choice technique for elective Caesarean section as simple, quick, reliable and cheap. However, this anaesthetic method can be burdened by maternal hypotension with significant maternal and foetal implications.

DETAILED DESCRIPTION:
Hypotension induced by neuraxial anaesthesia (NA-induced hypotension) is defined as systolic blood pressure (SBP) less than 100 mmHg or a decrease of 20-30% from baseline values. The incidence of hypotension could exceed 71% and can cause, if serious and prolonged, nausea, vomiting, lost of consciousness, placental hypoperfusion and foetal acidosis.

There are two alternative hypotheses to explain why hypotension might be so commonly diagnosed after regional analgesia during labour: preload reduction theory and afterload reduction theory. A non-invasive continue haemodynamic monitoring could be useful in detecting pregnant women with a positive preoperative supine stress, at increased risk for clinically significant hypotension during Caesarean section under spinal anaesthesia. These women seem more likely to benefit from optimizing the administration of fluids and vasoconstrictors to maintain pressure and cardiac output at basal levels.

Predictors of clinical need of therapy to counteract symptomatic hypotension (dependant variable) will be sought by using regression logistic analysis. Putative variable to include in the model will be selected through clinical and statistical criteria. Univariate screening will be performed assuming the usual cut-off of p<0,1 and taking into account the biological relevance. The final variable to challenge in the multivariate model will be selected according to the parsimony criteria in order to avoid overfitting and multicollinearity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with high bleeding risk (previous caesarean section, previous uterine surgery, placenta praevia/accrete, previous documented uterine atony, foetal macrosomia, polyhydramnios)
* Obstetric nulliparous or multiparous patients
* Spontaneous pregnancy
* Single foetus, at term
* Elective Caesarean section, fasting according to international guidelines
* At term BMI > 18 and < 35 kg/m2

Exclusion Criteria:

* Contraindications to neuraxial anaesthesia
* Previous documented maternal cardiovascular problems
* Gestational hypertension (defined as new onset systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg on two occasions at east 4 - 6 hours apart while the patient is on bed rest, with an appropriately sized cuff, after 20 weeks gestation)
* Chronic hypertension of any causes (defined as systemic blood pressure > 140/90 mmHg)
* Preeclampsia (defined as gestational hypertension with one or more of the following de novo conditions:

  * Proteinuria (defined as the excretion of 300 mg or more of protein in a 24-hour urine collection or a protein/creatinine ratio of at least 0.3 (each measured as mg/dL) or at least 1 g/L [2+] on dipstick testing)
  * Other maternal organ dysfunction:

    1. progressive renal insufficiency (renal creatinine concentration greater than 1.1 mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease),
    2. impaired liver function as indicated by abnormally elevated blood concentrations of liver enzymes (at least twice upper limit of normal concentration), severe persistent right upper quadrant or epigastric pain unresponsive to medication and not accounted for by alternative diagnoses, or both),
    3. new-onset cerebral or visual disturbances (examples include eclampsia, altered mental status, blindness, stroke, or more commonly hyperreflexia when accompanied by clonus, severe headaches when accompanied by hyperreflexia, persistent visual scotoma),
    4. haematological complications (thrombocytopenia - platelet count below 150,000/dL, disseminated intravascular coagulation (DIC), haemolysis).
* Uteroplacental dysfunction with foetal growth restriction (less than fifth percentile)
* Reversed end-diastolic flow on umbilical artery Doppler studies (IR > 0,5 at 24 week gestation)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy pregnant women admitted in the enrolling Centre to undergo to elective Caesarean section under spinal anaesthesia
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Stress tests and Systolic blood pressure | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Systolic blood pressure in mmHg) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Diastolic blood pressure | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Diastolic blood pressure in mmHg) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Mean arterial blood pressure | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Mean arterial blood pressure in mmHg) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Heart rate | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Heart rate in beats per minute) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Cardiac output | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Cardiac output in L/min) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Stroke volume | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Stroke volume in mL/beat) and neuraxial anaesthesia induced hypotension (clinical end point)
Stress tests and Systemic vascular resistance | before Caesarean section
  to identify correlations among stress tests (supine, deep breath in supine, left lateral, deep breath in left lateral, standing, deep breath in standing, leg raising), non-invasive haemodynamic parameter detected (Systemic vascular resistance in dynes - sec/cm^5) and neuraxial anaesthesia induced hypotension (clinical end point)

SECONDARY OUTCOMES:
Neuraxial induced hypotension | from immediately after induction of spinal anaesthesia to 15 minutes later
  Neuraxial induced hypotension is defined as a reduction of SBP < 100 mmHg or a decrease by 20 - 30%, compared to basal value

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Viviani, M.D., Principal Investigator — ASST Papa Giovanni XXIII, Bergamo, Italy
Locations (1):
- Asst Papa Giovanni Xxiii, Bergamo, Italy